CLINICAL TRIAL: NCT07260773
Title: The Effects of Coenzyme Q10 Pretreatment on Ovarian Function and Assisted Reproductive Outcomes in Patients With Poor Ovarian Response: A Single-Center Randomized Controlled Trial
Brief Title: The Effects of Coenzyme Q10 Pretreatment on Ovarian Function and Assisted Reproductive Outcomes in Patients With Ovarian Hyporesponsiveness.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Xiaohong Wang, Director of Obstetrics and Gynecology, Tangdu Hospital, Air Force Medical University Director of the Reproductive Medicine Center, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202507-08
Record Dates: First submitted 2025-09-30; First posted 2025-12-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Response
Keywords: Ovarian function
MeSH Terms: interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guidelines for Routine Treatment + Coenzyme Q10 (Experimental): Guidelines for Routine Treatment + Coenzyme Q10 (Nengqi Lang, Yunda Pharmaceutical) 30mg orally, 3 times daily, with pretreatment lasting 8 weeks. • ART treatment (in vitro fertilization (IVF)) commences during the first menstrual cycle following completion of treatment.
  Interventions: Dietary Supplement: Coenzyme Q10
- Guidelines for Routine Treatment plus placebo (Placebo Comparator): Guidelines for Routine Treatment plus placebo, administered for 8 weeks. ART treatment (IVF) commenced during the first menstrual cycle following completion of the treatment.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — One group received coenzyme Q10 pretreatment, while the other group did not. Following an 8-week pretreatment period, IVF cycles were performed, with regular follow-up evaluations conducted.
  Arms: Guidelines for Routine Treatment + Coenzyme Q10
Dietary Supplement: Placebo — Drug A plus placebo, administered for 8 weeks. ART treatment (IVF) commenced during the first menstrual cycle following completion of the treatment.
  Arms: Guidelines for Routine Treatment plus placebo

SUMMARY:
This prospective, randomized, double-blind, controlled study will be conducted at Tangdu Hospital, Air Force Medical University. It plans to enroll 128 patients with poor ovarian response for a 2-year study. The primary objective is to investigate the effects of exogenous coenzyme Q10 supplementation as pre-treatment on ovarian function and assisted reproductive clinical outcomes in patients with poor ovarian response.

Study Hypothesis: Coenzyme Q10 therapy is expected to effectively enhance ovarian function and improve assisted reproductive outcomes in patients with poor ovarian response, while demonstrating favorable safety profiles.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double-blind, controlled clinical trial designed to investigate the effects of coenzyme Q10 pretreatment on ovarian function and assisted reproductive clinical outcomes in patients with poor ovarian response (POR). The study will be conducted at Tangdu Hospital, Air Force Medical University, with an anticipated enrollment of 128 patients meeting the Bologna diagnostic criteria for POR. Participants will be randomly assigned to either the study group (Coenzyme Q10 group) or the control group (placebo group), with 64 patients in each group.

Study Group: Guidelines for Routine Treatment + Coenzyme Q10 (Nengqilang, Yuanda Pharmaceutical) 30mg orally, 3 times/day, for 8 weeks of pretreatment. ART treatment (in vitro fertilization (IVF)) commenced in the first menstrual cycle following completion of pretreatment.

Control Group: Guidelines for Routine Treatment + placebo for 8 weeks. ART (IVF) initiated in the first menstrual cycle following treatment completion.

Primary endpoints included oocyte retrieval rate and MII oocyte rate. Secondary endpoints encompassed total GnRHA dose, stimulation duration, peak E2 level, cycle cancellation rate, fertilization rate, high-quality embryo rate, clinical pregnancy rate, and miscarriage rate. Safety was assessed by adverse reaction incidence.

The study aims to validate the efficacy and safety of Coenzyme Q10 in improving ovarian response and ART outcomes in patients with poor ovarian response through scientifically rigorous design and statistical analysis. This will provide reliable evidence-based medical support for clinical practice and contribute to enhancing women's reproductive health.

ELIGIBILITY:
Inclusion Criteria:

* Individuals seeking IVF-ET fertility treatment;
* Meeting the Bologna criteria for the definition of poor ovarian response (POR), specifically:
* (1) Meeting 2 of the following 3 criteria:
* ① Presence of high-risk factors for POR;
* ② Previous cycle with ≤3 retrieved oocytes under a standard stimulation protocol;
* ③ Abnormal ovarian reserve assessment: Antral follicle count (AFC) <5 or Anti-Müllerian hormone (AMH) <1.1 ng/mL.

or

* (2) Patients with normal age or ovarian reserve function who experience poor ovarian response (POR) after two consecutive cycles of maximum ovarian stimulation protocols;
* BMI between 18.5-28.0 kg/m²
* Voluntarily participate and sign an informed consent form.

Exclusion Criteria:

* Age ≥40 years;
* Baseline FSH >25 U/L;
* Endocrine disorders (e.g., diabetes, thyroid disease) or autoimmune diseases (e.g., rheumatoid arthritis, lupus, Crohn's disease), chromosomal abnormalities, uterine malformations;
* History of ovarian surgery; history of uterine surgery; adenomyosis;
* History of more than 3 cycles of controlled ovarian stimulation (COS);
* Male infertility;
* Use within the past 3 months of medications that may affect ovarian reserve or ovarian responsiveness (e.g., oral contraceptives, glucocorticoids, antioxidant supplements, insulin sensitizers, DHEA, growth hormone, etc.);
* Use of traditional Chinese medicine within the past 3 months;
* Known allergy to Coenzyme Q10 or panthenol (water-soluble isomer of CoQ10);
* PGT (Preimplantation Genetic Testing) population;
* Acute or chronic renal insufficiency, hemodialysis treatment, history of severe renal impairment;
* Infectious diseases such as HIV, active hepatitis, history of metabolic acidosis, tuberculosis;
* Cardiovascular events within 3 months: coronary artery disease/myocardial infarction/clinically significant congestive heart failure; stroke/transient ischemic attack; deep vein thrombosis/pulmonary embolism; uncontrolled hypertension (systolic ≥160 mmHg or diastolic ≥90 mmHg); diagnosed diabetes; coronary intervention or coronary artery bypass graft surgery;
* Neurological disorders such as dementia (e.g., Alzheimer's/Parkinson's) or use of related medications;
* History of psychological/psychiatric disorders and use of antiepileptic, antidepressant, or similar medications;
* History of cancer, radiation therapy, or chemotherapy;
* Unwillingness to take supplements provided by this study;
* Alcoholics, smokers, or individuals with substance dependence;
* Participants in other clinical trials within the past month;
* Patients deemed ineligible for enrollment by the investigator.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 128 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | From the start of pretreatment until the IVF oocyte retrieval day (approximately 8 weeks of pretreatment plus one IVF treatment cycle).
  Total number of oocytes retrieved during the oocyte retrieval procedure(unit: count).
Rate of Metaphase II (MII) Oocytes | From the start of pretreatment until the IVF oocyte retrieval day (approximately 8 weeks of pretreatment plus one IVF treatment cycle).
  The proportion of mature oocytes (Metaphase II oocytes) among the total number of oocytes retrieved (unit: percentage).

SECONDARY OUTCOMES:
Total Gonadotropin (Gn) Dose | From the start of ovarian stimulation until the HCG trigger day (up to approximately 2 weeks).
  Total dosage of Gonadotropin (Gn) used during one IVF stimulation cycle (unit: International Units, IU).
Days of stimulation | From the start of ovarian stimulation until the HCG trigger day (up to approximately 2 weeks).
  Total number of days from the initiation of Gonadotropin (Gn) to the HCG trigger day in one IVF cycle (unit: days).
Peak Estradiol (E2) Level | Assessed on the HCG trigger 1 day.
  Serum estradiol level measured on the day of HCG trigger (unit: pg/mL).
Cycle Cancellation Rate | From the start of ovarian stimulation until the scheduled oocyte retrieval day (up to approximately 2 weeks).
  The proportion of cycles cancelled due to poor ovarian response (e.g., inadequate follicular development) without proceeding to oocyte retrieval (unit: percentage).
Fertilization rate | Day 1 after oocyte retrieval (fertilization assessment)
  The percentage of fertilized oocytes out of the total number of retrieved oocytes.
Normal fertilization rate | Day 1 after oocyte retrieval (fertilization assessment)
  The percentage of fertilized oocytes with two pronuclei (2PN) out of the total fertilized oocytes.
Cleavage Rate | Day 3 after oocyte retrieval (embryo development assessment)
  The percentage of fertilized oocytes that undergo cleavage out of the total fertilized oocytes.
Day 3 High-Quality Embryo Rate | Day 3 after oocyte retrieval (embryo morphology scoring)
  The percentage of high-quality embryos on Day 3 out of all Day 3 embryos.
Clinical Pregnancy Rate (First Transfer Cycle) | From pretreatment initiation until 6 weeks after the first embryo transfer.
  The percentage of cycles with a gestational sac and fetal cardiac activity observed via transvaginal ultrasound approximately 5 weeks after the first embryo transfer, out of the total number of first transfer cycles.
Miscarriage Rate | From confirmation of clinical pregnancy until 20 weeks of gestation.
  The percentage of cycles with pregnancy loss after clinical confirmation of pregnancy out of all clinically pregnant cycles.

OTHER OUTCOMES:
Incidence of Adverse Reactions | From the first dose of the study drug until 6 weeks after the first embryo transfer (for clinical pregnancy assessment).
  The incidence of adverse events occurring during the treatment period.

IPD SHARING:
Plan to Share IPD: No